CLINICAL TRIAL: NCT05206253
Title: Egg Versus Whey Protein as the Optimal Supplement for Fitness-conscious People
Brief Title: Effectiveness of Egg Versus Whey Protein Powder During Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Egg Farmers of Canada (Unknown)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Bio 2962
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole egg powder (Experimental): Dietary supplementation with whole egg powder after resistance training sessions
  Interventions: Dietary Supplement: Whole egg powder
- Whey protein powder (Active Comparator): Dietary supplementation with whey protein powder after resistance training sessions
  Interventions: Dietary Supplement: Whey protein powder
- Maltodextrin placebo (Placebo Comparator): Dietary supplementation with maltodextrin placebo after resistance training sessions
  Interventions: Dietary Supplement: Maltodextrin placebo

INTERVENTIONS:
Dietary Supplement: Whole egg powder — Nutritional supplementation during a 12 week resistance training program
  Arms: Whole egg powder
Dietary Supplement: Whey protein powder — Nutritional supplementation during a 12 week resistance training program
  Arms: Whey protein powder
Dietary Supplement: Maltodextrin placebo — Nutritional supplementation during a 12 week resistance training program
  Arms: Maltodextrin placebo

SUMMARY:
Consumption of whole eggs has recently been shown to stimulate muscle protein synthesis to a greater degree than consumption of egg whites after a resistance training session. It is theorized that the egg yoke contains bio-active nutrients that enhance the protein provided by egg whites. The study will evaluate the effect of whole egg powder compared to whey protein powder and placebo over 12 weeks of resistance training in men and women who are participating in resistance training programs.

DETAILED DESCRIPTION:
Consuming whole eggs after resistance training sessions appears to be more effective for simulating muscle protein synthesis that simply consuming egg whites. The egg yolks might enhance the effect of protein derived from egg whites. The study will compare post-exercise supplementation with about 30 grams of protein derived from whole egg powder versus whey protein powder and placebo (maltodextrin) over a 12-week resistance training program. Resistance-trained men and women (n=120) will be randomized to consume either the whole-egg powder, whey protein powder or maltodextrin after resistance training 6 times per week for 12 weeks. The primary outcome measure is change in lean tissue mass. Secondary measures include change in fat mass, change in arm and leg muscle thickness, change in bench press, squat, and knee extension strength, and change in fasting blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Resistance training experience for at least one year

Exclusion Criteria:

* Having taken any nutritional supplements the past 30 days
* Currently using anabolic steroids
* Currently taking corticosteroids
* Allergies to dairy or egg products
* Identifying any medical conditions as determined by the "Get Active Questionnaire"

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in lean tissue mass | 12 weeks
  Lean tissue mass measured by DXA

SECONDARY OUTCOMES:
Change in fat mass | 12 weeks
  Fat mass measured by DXA
Change in biceps muscle thickness | 12 weeks
  biceps muscle thickness measured by ultrasound
Change in triceps muscle thickness | 12 weeks
  triceps muscle thickness measured by ultrasound
Change in quadriceps muscle thickness | 12 weeks
  quadriceps muscle thickness measured by ultrasound
Change in hamstrings muscle thickness | 12 weeks
  hamstrings muscle thickness measured by ultrasound
Change in bench press strength | 12 weeks
  Bench press strength (kg)
Change in leg squat strength | 12 weeks
  Leg squat strength (kg)
Change in knee extension strength | 12 weeks
  Isokinetic knee extension torque
Change in fasting glucose | 12 weeks
  Fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan; Darren Candow, Ph.D., Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - University of Regina, Regina, Saskatchewan
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No